CLINICAL TRIAL: NCT04492917
Title: The Effect of CV4 and Sacral Technique on the Alpha Bands Power: A Randomized Controlled Trial
Brief Title: The Effect of CV4 and Sacral Technique on the Alpha Bands Power
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Superiore di Osteopatia di Milano (Other)
Responsible Party: Principal Investigator, Viviana Pisa, Principal Investigator, Istituto Superiore di Osteopatia di Milano
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CV4 Alpha Band
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Healthy; Osteopathic Manipulation
Keywords: EEG; Alpha Rhythm; CV4

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranial Technique CV4 (Experimental): All subjects received a combination of the active technique (CV4) and the corresponding sham technique (shamCV4).
  CV4: the lateral angles of the occipital squama are manually approximated slightly exaggerating the posterior convexity of the occiput and taking the cranium into sustained extension. The technique ended when the osteopath perceived the still point, a condition in which the balanced membranous or ligamentous tension is achieved.
  ShamCV4: sham intervention was performed by placing the hands in the same position as the corresponding active technique, applying a light touch
  Interventions: Other: CV4; Other: Sham CV4
- Sacral Technique ST (Active Comparator): All subjects received a combination of the active technique (ST) and the corresponding sham technique (sST).
  ST: The subject was lying in the supine position, while the osteopath positioned the index and middle fingers of the caudal hand on either side of the subject's sacrum. Then establishes a point of balance between the coccyx and the vertex facilitating the sacral extension until the achievement of the still point.
  ShamST: sham intervention was performed by placing the hands in the same position of the corresponding active technique, applying a light touch
  Interventions: Other: ST; Other: Sham ST

INTERVENTIONS:
Other: CV4 — The osteopath was sitting at the head of the examination table, with the subject lying supine. The osteopath approximated with the hands the lateral angles of the occipital squama, taking the cranium into sustained extension. The technique ended when the osteopath perceived the still point, a condition in which the balanced membranous or ligamentous tension is achieved.
  Arms: Cranial Technique CV4
Other: ST — The subject was lying in the supine position, while the osteopath positioned the index and middle fingers of the caudal hand on either side of the subject's sacrum. Then establishes a point of balance between the coccyx and the vertex facilitating the sacral extension until the achievement of the still point
  Arms: Sacral Technique ST
Other: Sham CV4 — the sham intervention was performed by placing the hands in the same position as the corresponding active technique, applying a light touch
  Arms: Cranial Technique CV4
Other: Sham ST — The sham intervention was performed by placing the hands in the same position as the corresponding active technique, applying a light touch
  Arms: Sacral Technique ST

SUMMARY:
Compression of the fourth ventricle (CV4), is the most studied cranial technique, commonly used by Osteopathy in Cranial Field practitioners. Evidence attributed to CV4 some effects on nervous system functions, however, the supporting evidence for CV4 clinical benefits is promising but still poor. The osteopathic tradition considers the sacrum linked to the cranium through anatomical and functional connections. To our knowledge, no studies explored the potential effect of a sacral technique on brain activity as an indicator of a neurophysiological connection between the occiput and sacrum. This study aims to explore this effect by measuring the alpha-band activity during the application of a sacral technique (ST) compared to the CV4 application.

DETAILED DESCRIPTION:
Forty healthy volunteers will receive a combination of CV4 technique, CV4 sham, sacral technique (ST) and sacral sham technique (sST).

Each session, split by a 4-hour washout, will start with 10 min of no treatment (resting state), followed by two randomized interventions. Alpha EEG will be continuously recorded during each intervention and 10 min after, for a total of approximately 50-60 min per session.

ELIGIBILITY:
Inclusion Criteria:

* Age
* Subjects had to sleep for at least 6 hours the night before the experiment

Exclusion Criteria:

* Use of Psychoactive or Psychotropic Substances
* Cerebrovascular diseases
* Recent headaches
* Use of nicotine in the 24 hours prior to the quantitative EEG registration
* Use of alcohol in the previous 12 hours.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Alpha EEG | 50 minutes
  Quantitative EEG recording of alpha wave (8-12Hz)

CONTACTS AND LOCATIONS:
Overall Officials: Pisa, Principal Investigator — Istituto Superiore di Osteopatia
Locations (1):
- Centro di Medicina Osteopatica, Milan, Italy

IPD SHARING:
Plan to Share IPD: No